CLINICAL TRIAL: NCT02036294
Title: An Integrative Multilevel Study for Improving Patient-Centered Care Delivery Among Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Improving Patient-Centered Care Delivery Among Patients With Chronic Obstructive Pulmonary Disease
Acronym: BREATHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00090518; IH-1304-7118 (Other: Other)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Patient self-care behaviors; Patient activation; Family caregiver support; Patient-centered care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Participation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other): Usual Care: Standard healthcare services will be received. Study participants in this arm will not receive any additional study interventions.
  Interventions: Other: Usual Care
- BREATHE program (Experimental): Study participants randomized to this arm will be offered the BREATHE program an integrated multifaceted intervention that includes comprehensive biopsychosocial assessment, a tailored treatment plan, a tailored disease management program, and care management support services .
  Interventions: Other: BREATHE program

INTERVENTIONS:
Other: BREATHE program — A patient and family- centered transitional care intervention that includes a comprehensive biopsychosocial assessment, a tailored treatment plan, a tailored disease management program, and care management support services .
  Arms: BREATHE program
Other: Usual Care — Standard Healthcare Services
  Arms: Usual Care

SUMMARY:
This study involves development and testing of a patient and family-centered transitional care program for patients who are hospitalized with Chronic Obstructive Pulmonary Disease (COPD) exacerbations. The study intervention includes tailored services to address individual patients' biopsychosocial needs, starting early during hospital stay and continuing for 3 months post hospital discharge.

The study hypothesis is that compared to usual care, the study intervention will : a) Improve patient health- related quality of life and survival, and reduce use of hospital and emergency room visits; b) result in improved patient experience, self- confidence, and self-care behaviors; c) result in improved family caregivers coping skills, self-confidence, and problem solving skills to address patient barriers to care and treatment.

DETAILED DESCRIPTION:
This study evaluates using a randomized controlled trial design the impact of a patient and family-centered transitional care program named the BREATHE program. The BREATHE program stands for 'Better Respiratory Education and Treatment Help Empower'. The BREATHE program offers the following:

1. Individualized transition support services to help ensure that the patient (and family caregiver if available) are prepared for discharge, understand the discharge plan of care, and receive post discharge follow up to help meet their needs
2. Tailored COPD self-management education and support program that starts during the hospital stay and continues post discharge in the community setting
3. Facilitated access to community based services.

The intervention is delivered by a new team member called "COPD Nurse Transition Guide". The new team member works with both the hospital and outpatient care teams, is a registered nurse with homecare services experience, and have received additional training in COPD self-management and motivational interviewing. The nurse meets participants in the hospital and then follows up with them via home visits and phone calls.The intervention involves both patients and family caregivers (if available), is literacy adapted, and follows a tailored approach based on patient needs, priorities, and preferences.

ELIGIBILITY:
Inclusion criteria:

* Admitted to the hospital with a diagnosis of an acute COPD exacerbation; OR has a previous COPD diagnosis* AND receiving treatment to control COPD symptoms - (e.g. nebulizer treatment, prednisone course, …) in the current hospitalization
* Age > 40 and >10 pack-yrs smoking
* English speaking
* Anticipated discharge back to home (rather than to Hospice or long term nursing home placement)

Exclusion criteria:

* Severe cognitive dysfunction
* Terminal illness (less than 6 months life expectancy) that is non-COPD related
* Homeless (no home address)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Aboumatar, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Aboumatar H, Naqibuddin M, Chung S, Chaudhry H, Kim SW, Saunders J, Bone L, Gurses AP, Knowlton A, Pronovost P, Putcha N, Rand C, Roter D, Sylvester C, Thompson C, Wolff JL, Hibbard J, Wise RA. Effect of a Hospital-Initiated Program Combining Transitional Care and Long-term Self-management Support on Outcomes of Patients Hospitalized With Chronic Obstructive Pulmonary Disease: A Randomized Clinical Trial. JAMA. 2019 Oct 8;322(14):1371-1380. doi: 10.1001/jama.2019.11982. PMID 31593271
- [Derived] Aboumatar H, Naqibuddin M, Chung S, Chaudhry H, Kim SW, Saunders J, Bone L, Gurses AP, Knowlton A, Pronovost P, Putcha N, Rand C, Roter D, Sylvester C, Thompson C, Wolff JL, Hibbard J, Wise RA. Effect of a Program Combining Transitional Care and Long-term Self-management Support on Outcomes of Hospitalized Patients With Chronic Obstructive Pulmonary Disease: A Randomized Clinical Trial. JAMA. 2018 Dec 11;320(22):2335-2343. doi: 10.1001/jama.2018.17933. PMID 30419103 (Retraction: PMID 31593277 JAMA. 2019 Oct 8;322(14):1417-1418)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | BREATHE Program
Started | 120 | 120
Completed | 111 | 109
Not Completed | 9 | 11
Not completed — Death | 7 | 8
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | BREATHE Program | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (10.0) | 63.9 (9.6) | 64.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 72 | 148
  Male | 44 | 48 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 116 | 116 | 232
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 20 | 38
  White | 100 | 98 | 198
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Total score of St. George's Respiratory Questionnaire (SGRQ) [Mean (Standard Deviation); unit: units on a scale] — St. George's Respiratory Questionnaire (SGRQ) is a validated instrument to measure the health-related quality of life among patients with respiratory disease. The total score range is 0 to 100, with 0 representing best score and 100 worst score. Average of scores (with standard deviation) for participants in each arm is reported.
  units on a scale | 63.6 (17.4) | 62.3 (18.8) | 62.9 (19.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Chronic Obstructive Pulmonary Disease (COPD)-Related Hospitalizations and Emergency Department (ED) Visits Per Patient Within Each Study Arm
Description: The primary outcome measure in this study is the mean number of COPD-related hospitalizations and ED visits per patient within each study arm . The number of hospital and ED visits per patient were counted at 6 months post 'index-hospitalization'. Index-hospitalization refers to the hospitalization in which the patient was enrolled into the study. A COPD- related hospitalization was defined as a hospitalization with discharge diagnosis of COPD exacerbation or Pneumonia; a hospitalization where the participant was admitted for congestive heart failure but received treatment for COPD exacerbation (nebulizer treatment plus steroids) ; or, admitted for symptoms pertaining to COPD and received steroids. A COPD- related ED visit was defined as a visit where the treating physician stated that the visit reason is COPD; or, where the participant was discharged on treatment with oral steroids or on treatment for pneumonia.
Time Frame: Measured at 6 months post 'index-hospitalization'
Population: Data was analyzed for all participants unless: 1) participant died during the 6 months study period (we have to exclude deaths from this analysis because we cannot calculate a full count of hospital or ED visits during the 6 months period if the participant had died before the 6 months has elapsed ) ; 2) participant withdrew from the study.
Measure: Mean (Standard Deviation); unit: COPD-related visits per participant
Arm/Group | Usual Care | BREATHE Program
Number analyzed (Participants) | 113 | 112
COPD-related visits per participant | 0.72 (1.38) | 1.40 (2.08)

2. Primary Outcome: Mean Change in Patients' Score on the St. George Respiratory Questionnaire Within Each Study Arm
Description: This outcome measures the mean change in patient participants' quality of life as measured by the Saint George's Respiratory Questionnaire (SGRQ) score over the 6 month study period within each study arm.The St. George Respiratory Questionnaire (SGRQ) is a widely used validated disease- specific instrument that measures health-related quality of life. The SGRQ measures, using patient self-report, disease impact on symptoms, patient activity, and daily life. The total score for SGRQ ranges from 0 to 100, with higher scores indicating more limitations. The change in a patient's quality of life was calculated as the difference in their total score at 6 months post index-hospitalization from baseline. A difference of 4 points in total score is considered a clinically meaningful difference.
Time Frame: Baseline to 6 months post index-hospitalization
Population: Not all participants could be reached to complete the survey
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | BREATHE Program
Number analyzed (Participants) | 91 | 88
units on a scale | -2.69 [-9.34 to 3.96] | 2.81 [-3.73 to 9.34]

3. Secondary Outcome: Mean Number of Chronic Obstructive Pulmonary Disease (COPD)-Related Hospitalizations and Emergency Department (ED) Visits Per Patient Within Each Study Arm
Description: The primary outcome measure in this study is the mean number of COPD-related hospitalizations and ED visits per patient within each study arm . The number of hospital and ED visits per patient were counted at 1 month post 'index-hospitalization'. Index-hospitalization refers to the hospitalization in which the patient was enrolled into the study. A COPD- related hospitalization was defined as a hospitalization with discharge diagnosis of COPD exacerbation or Pneumonia; a hospitalization where the participant was admitted for congestive heart failure but received treatment for COPD exacerbation (nebulizer treatment plus steroids) ; or, admitted for symptoms pertaining to COPD and received steroids. A COPD- related ED visit was defined as a visit where the treating physician stated that the visit reason is COPD; or, where the participant was discharged on treatment with oral steroids or on treatment for pneumonia.
Time Frame: Measured at 1 month post 'index-hospitalization'
Population: Data was analyzed for all participants unless: 1) participant died during the 1 month study period (we have to exclude deaths from this analysis because we cannot calculate a full count of hospital or ED visits during the 1 month period if the participant had died before the 1 month have elapsed ) ; 2) participant withdrew from the study.
Measure: Mean (Standard Deviation); unit: COPD-related visits per participant
Arm/Group | Usual Care | BREATHE Program
Number analyzed (Participants) | 119 | 118
COPD-related visits per participant | 0.12 (0.32) | 0.27 (0.59)

4. Secondary Outcome: Mean Number of Chronic Obstructive Pulmonary Disease (COPD)-Related Hospitalizations and Emergency Department (ED) Visits Per Patient Within Each Study Arm
Description: The primary outcome measure in this study is the mean number of COPD-related hospitalizations and ED visits per patient within each study arm. The number of hospital and ED visits per patient were counted at 3 months post 'index-hospitalization'. Index-hospitalization refers to the hospitalization in which the patient was enrolled into the study. A COPD- related hospitalization was defined as a hospitalization with discharge diagnosis of COPD exacerbation or Pneumonia; a hospitalization where the participant was admitted for congestive heart failure but received treatment for COPD exacerbation (nebulizer treatment plus steroids) ; or, admitted for symptoms pertaining to COPD and received steroids. A COPD- related ED visit was defined as a visit where the treating physician stated that the visit reason is COPD; or, where the participant was discharged on treatment with oral steroids or on treatment for pneumonia.
Time Frame: Measured at 3 months post 'index-hospitalization'
Population: Data was analyzed for all participants unless: 1) participant died during the 3 months study period (we have to exclude deaths from this analysis because we cannot calculate a full count of hospital or ED visits during the 3 months period if the participant had died before the 3 months have elapsed ) ; 2) participant withdrew from the study.
Measure: Mean (Standard Deviation); unit: COPD-related visits per participant
Arm/Group | Usual Care | BREATHE Program
Number analyzed (Participants) | 115 | 116
COPD-related visits per participant | 0.43 (0.90) | 0.78 (1.24)

5. Secondary Outcome: Mean Change in Patients' Score on the St. George Respiratory Questionnaire Within Each Study Arm
Description: This outcome measures the mean change in patient participants' quality of life as measured by the Saint George's Respiratory Questionnaire (SGRQ) score over the 3 month study period within each study arm.The St. George Respiratory Questionnaire (SGRQ) is a widely used validated disease- specific instrument that measures health-related quality of life. The SGRQ measures, using patient self-report, disease impact on symptoms, patient activity, and daily life. The total score for SGRQ ranges from 0 to 100, with higher scores indicating more limitations. The change in a patient's quality of life was calculated as the difference in their total score at 3 months post index-hospitalization from baseline. A difference of 4 points in total score is considered a clinically meaningful difference.
Time Frame: Baseline to 3 months post index-hospitalization
Population: Not all participants could be reached to complete the survey
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | BREATHE Program
Number analyzed (Participants) | 90 | 82
units on a scale | -1.13 (17.14) | -0.85 (19.44)

6. Secondary Outcome: Probability for Survival Without Death or a COPD- Related Acute Care Event at 6 Months Post Index-hospitalization, Estimated Using the Kaplan-Meier Method
Description: Kaplan-Meier probability estimates that a participant would have their first event (death or COPD- related hospitalization or ED visit) sometime after 6 months from their index- hospitalization. The estimates are provided as the proportion of participants who do not have an event at 6 months post their index hospitalization.
Time Frame: Measured at 180 days post-discharge from index hospitalization
Population: All participants whose medical records were available to confirm whether a hospitalization or ED visit is COPD-related
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Usual Care | BREATHE Program
Number analyzed (Participants) | 120 | 119
Proportion of participants | 0.58 [0.49 to 0.66] | 0.45 [0.35 to 0.53]

ADVERSE EVENTS:
Time Frame: Between study enrollment and 6 months
Description: Deaths were assessed systematically via medical records and vital statistics records review.
  All hospitalization events were assessed systematically via patient report and medical records review.
  Other serious adverse events voluntarily reported by patient or nurse
Arm/Group | Usual Care | BREATHE Program
All-Cause Mortality (participants affected / at risk) | 7/120 | 8/120
Serious Adverse Events (participants affected / at risk) | 69/120 | 76/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=120) | BREATHE Program (N=120)
Hospitalization for any cause (General disorders) | 69 (137) | 76 (202) — These events are hospitalizations of any cause that occurred during the study period (between study enrollment and 6 months). These are anticipated adverse events.
Other serious unanticipated events (General disorders) | 0 (0) | 0 (0) — Event voluntarily reported by patient or nurse

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes